CLINICAL TRIAL: NCT07264309
Title: Combined Intravenous Tramadol and Paracetamol Versus Intramuscular Pethidine for Pain Relief During the First Stage of Labor
Brief Title: Combined Intravenous Tramadol and Paracetamol Versus Intramuscular Pethidine for Pain Relief During the First Stage of Labor. Compare the Efficacy and Adverse Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zohar Nachum (Other)
Responsible Party: Sponsor-Investigator, Zohar Nachum, Professor, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37-24
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2024-12

CONDITIONS: Pain Management; Birth
MeSH Terms: conditions — Agnosia | interventions — Meperidine; Tramadol; Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of paracetamol and tramadol (Experimental): Women will receive intravenous infusion of 50 ml contain 1000mg paracetamol and 100ml contain 100mg tramadol over 15 min
  Interventions: Drug: Tramadol; Drug: Paracetamol 1 g
- Pethidine (Active Comparator): 75 mg of pethidine will be given intramuscularly in the upper - outer quadrant of the
  Interventions: Drug: pethidine

INTERVENTIONS:
Drug: pethidine — 75 mg of pethidine will be given intramuscularly in the upper - outer quadrant of the
  Arms: Pethidine
Drug: Tramadol — Women will receive intravenous infusion of 100 ml containing 100 mg of tramadol over 15 min
  Arms: Combination of paracetamol and tramadol
Drug: Paracetamol 1 g — women will receive 50 ml containing 1000 mg of paracetamol IV over 15 min
  Arms: Combination of paracetamol and tramadol

SUMMARY:
The goal of this intervention study is to compare the efficacy and adverse effects of pain relief during the first stage of labor using 75 mg IM pethidine versus the combination of IV 100 mg tramadol and 1000 mg paracetamol.

The investigator assume that the combination of IV tramadol and paracetamol will be more effective with less adverse effects than IM pethidine in pain relief at the first stage of labor.

The investigator primary outcome is The effect on pain relief according to numeric rating scale (NTS) in the study groups Before the administration of the drugs, fetal heart rate patterns and contractions will be recorded with cardiotocography monitor for at least 20 min. The investigator will evaluate vigilance at 30 minutes following drug administration.

NRS pain score (0-10) will be collected before administration and one hour after drug administration

ELIGIBILITY:
Inclusion Criteria:

Singleton Term pregnancy First stage of labor including at least 4 painful contractions in 30 min with cervical dilatation less or equal to 1 cm or 50% effacement Spontaneous or induced labor -

Exclusion Criteria:

* Previous cesarean delivery
* Malpresentation
* Multiple pregnancies
* Suspected intrauterine growth restriction < 3 percentile
* Suspected placental abruption
* History of allergy to paracetamol, tramadol or pethidine
* Women with sleep apnea disorder
* Morbid obesity BMI≥40
* History of significant cardiac, liver and renal diseases
* Anti-convulsive medication consumption
* MAO inhibitors medication consumption within the last 14 days
* Non reassuring fetal heart rate monitoring (type II or III)
* Tense use

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The effect on pain relief | one hour after drug administration.
  according to numeric rating scale (NRS), which runs from 0-10, where 0 is "no pain" and 10 is the "worst pain.

SECONDARY OUTCOMES:
Women satisfactory rate by NRS- a scale between 1-5, where 1 is no satisfactory and 5- is excellent satisfactory | from enrollment up to 72 hours after the birth
Maternal adverse effects of the medications | from enrollment to 72 hours after birth
First stage of labor duration (hours) | from enrollment to 72 hours after birth
The need for additional analgesia (Epidural, pethidine IV, nitrous) | from enrollment to 72 hours after birth
Fetal and neonatal outcomes | from enrollment to 72 hours after birth
Pregnancy outcomes | from birth up to 72 hours after birth

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek MC, Afula, Israel

IPD SHARING:
Plan to Share IPD: No